CLINICAL TRIAL: NCT03175055
Title: Phoenix Exoskeleton Clinical Study
Brief Title: Phoenix Exoskeleton for SCI Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10133
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Phoenix (Experimental): Phoenix
  Interventions: Device: Phoenix

INTERVENTIONS:
Device: Phoenix — The study to assess safety and efficacy of Phoenix medical exoskeleton.

SUMMARY:
This study will evaluate the Phoenix device for safety and effectiveness at allowing persons with SCI who are non-ambulatory or poorly ambulatory to stand up and walk under a variety of conditions.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years of age or older in general good health
2. Weigh no more than 220lbs
3. Skin must be healthy where it touches the Phoenix
4. Able to stand using a device such as a standing frame
5. Have enough strength in your hands and shoulders to support yourself standing and walking using crutches or a walker
6. Have good control of upper body
7. Determined to have enough bone health to walk full weight bearing without risk of fracture. Meeting of this condition is at the discretion of your personal MD
8. Passive range of motion (PROM) at shoulders, trunk, upper extremities and lower extremities within functional limits for safe gait and use of appropriate assistive device/stability aid
9. Hip width no greater than 18" (46 cm) measured when sitting.
10. Femur length between 12.3 inches (31.3 cm) and 19.8 inches (50.2 cm) measured between centers of hip and knee joints.
11. Tibia length between 13.4 inches (33.9 cm) and 22 (55.9 cm) inches measured between the knee joint and bottom of the foot.
12. In general good health and able to tolerate moderate levels of activity.
13. Blood pressure and heart rate within established guidelines for locomotive training:

At rest; Systolic 150 or less Diastolic 90 or less and Heart rate 100 or less Exercise; Systolic 180 or less Diastolic 105 or less and Heart Rate 145 or less

Exclusion Criteria:

* 1. Pregnant or lactating females 2. Spinal cord injury level higher than T4 3. Severe muscle stiffness/tightness 4. Significant spasticity (Modified Ashworth Scale score of 3 or above) 5. Trunk or lower extremity pressure ulcer 6. Open Wounds 7. Unstable spine, un-healed limbs, or fractures 8. Severe sensitivity to touch 9. Presence of bone in soft tissue where bone normally does not exist (heterotopic ossification), limiting range of motion in the hip or knee joints 10. Joint instability, dislocation, moderate to severe hip dysplasia 11. Significant scoliosis (>40 degrees) 12. Hardware, implant, or any external device impeding with safe fitting or use of Phoenix 13. Femoral or tibial rotation deformity (>15 degrees) 14. Significant flexion contractures limited to 35º at the hip and 20º at the knee 15. Uncontrolled seizures, musculoskeletal injury, fracture or lower-limb surgery in past year.

  16. Known history of pulmonary disease limiting exercise tolerance or history of cardiac disease 17. Psychopathology, or other condition that the physician or investigator, in his or her clinical judgment, considers to be exclusionary to safely use an exoskeleton.

  18. Severe concurrent medical diseases, illness, systemic or peripheral infection 19. Dizziness or headache with standing 20. History of autonomic dysreflexia 21. Orthostatic Hypotension: Decrease in Systolic BP > 20, Diastolic BP > 10 upon standing from a seated position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | 10 weeks
6 Minute Walk Test (6MWT) | 10 weeks
10 Meter Walk Test (10MWT) | 10 weeks

SECONDARY OUTCOMES:
Surface Walk Test | 10 weeks
  Testing the ability to ambulate with the device on a variety of surfaces

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - suitX, Emeryville, California
  - Motion & Gait Lab, Lucile Packard Children's Hospital Stanford, Menlo Park, California
  - St. David's Medical Center, Rehabilitation Hospital, Austin, Texas
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided